CLINICAL TRIAL: NCT06570447
Title: An Open-label, Single-arm, Single-center, Phase II Clinical Trial of Glofitamab Combination With Chidamide in Patients With Recurrent and Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Glofitamab Combination With Chidamide in Patients With Recurrent/Refractory DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Huilai Zhang, Director of lymphoma department, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTC-RR-DLBCL01
Record Dates: First submitted 2024-08-11; First posted 2024-08-26 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Diffuse Large B-Cell Lymphoma-Recurrent; Diffuse Large B-Cell Lymphoma-Refractory
MeSH Terms: interventions — glofitamab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination therapy of Glofitamab, chidamide (Experimental): Each subject will be given combination therapy of Glofitamab, chidamide. Glofitamab Injection with 2.5 mg on D8 and 10 mg on D15 in Cycle 1; with 30mg in Cycle 2-12, every 3 weeks.
  Interventions: Drug: Glofitamab; Drug: Chidamide

INTERVENTIONS:
Drug: Glofitamab — For Glofitamab Injection solution, after Obinutuzumab pretreatment on Day 1 of Cycle 1, patients followed a step-dose escalation regimen.
Drug: Chidamide — Chidamide: 30 mg/d orally twice a week for 21 days as a treatment cycle.

SUMMARY:
An open-label, single-arm, single-center, phase II clinical trial to evaluate the feasibility, efficacy and safety of Glofitamab Combination with chidamide in patients with recurrent/refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
This is an open-label, single-arm, single-center study to evaluate the feasibility, efficacy and safety of Glofitamab Combination with chidamide in the patient ≥ 18 years of age with recurrent/refractory diffuse large B-cell lymphoma. Subjects who meet the eligibility criteria will receive combination therapy of Glofitamab, chidamide. The study will include the following sequential phases: screening, treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

- To be eligible for enrollment in this study, a subject must meet all of the following criteria:

1. Signed informed consent
2. Age ≥ 18 years at the time of informed consent
3. Patients must be willing and able to comply with protocol-specified hospitalization requirements following administration of Glofitamab. Patients must also be willing to comply with all study-related procedures.
4. Histologically confirmed DLBCL, including any of the following 2016 WHO Lymphocytes Neoplasm classifications (Swerdlow et al. 2016) Diagnosis: DLBCL-NOS, HGBCL, PMBCL and FL transformed DLBCL (trFL)

   - A pathology report (if available) from the initial histopathological diagnosis must be provided. Patients with trFL must also provide a pathology report (if available) at the time of disease transformation. Results of all tissue tests performed at initial diagnosis should be provided, including but not limited to tests to assess cellular origin, BCL2, and MYC abnormalities (if performed).
5. Patients must have relapsed or Cap following at least two prior lines of systemic therapy (including at least one prior regimen containing anthracene Treatment failure and at least one prior regimen containing anti-CD20 targeted therapy).

   * Patients may have received Autologous haematopoietic stem cell transplant (HSCT) prior to recruitment; consolidative autologous HSCT after Chemotherapy will be counted as a line of therapy.
   * CAR T cells plus bridging were counted as a treatment line.
   * Local therapies (e.g., radiotherapy) will not be considered as treatment lines.
6. Patients must have measurable disease: at least one bidimensionally measurable Lymphadenopathy, defined as > 1.5 cm in the longest diameter; or at least one bidimensionally measurable extranodal lesion, defined as > 1.0 cm in the longest diameter.
7. Verify availability of Neoplasm tissues, unless not available per investigator assessment. Freshly collected Biopsy specimens are preferred. Representative Neoplasm tissue specimens or unstained serial sections are acceptable.
8. Eastern Cooperative Neoplasm Group (ECOG) performance status of 0 or 1
9. Life expectancy (as assessed by the investigator) ≥ 12 weeks
10. Carcinoma due to prior anti Adverse event therapy must have resolved to ≤ grade 1 (except Alopecia and Hyporexia).
11. Adequate liver function

    * Bilirubin total ≤ 1.5 x upper limit of normal (ULN); patients with documented history of Gilbert's syndrome: Bilirubin total ≤ 3 x ULN with elevated indirect Bilirubin;
    * AST/ALT ≤ 3 × ULN
12. Adequate hematological function:

    * Neutrophil count ≥ 1.5 x 109 cells/L (1.500/μL);
    * Platelet count ≥ 75,000/μL (and no Platelet transfusion within 14 days before Gpt administration on Day 1 of Cycle 1);
    * Haemoglobin ≥ 10.0 g/dL (6.2 mmol/L); no Transfusion within 21 days prior to Gpt dosing on Cycle 1 Day 1
13. Adequate renal function: Serum creatinine ≤ 1.5 × ULN or Creatinine clearance ≥ 50 mL/min calculated according to the C OC kroft Gault formula (see Appendix 14) (patients whose renal function is not adequately reflected by Serum creatinine levels as judged by the investigator)
14. Negative serum Pregnancy test within 7 days prior to study treatment for women of childbearing potential. Amenorrhoea is not required for women of non-childbearing potential who are post-menopausal (≥ 12 months of non-therapeutic Surgery) or Pregnancy test sterilized (absence of ovaries and/or uterus). For women of childbearing potential: Agree to remain abstinent (avoid heterosexual intercourse) or to take Contraception measures.
15. For men: Agree to remain abstinent (avoid heterosexual intercourse) or practice Contraception

Exclusion Criteria:

Any subject who meets any of the following criteria should not be enrolled in the study:

1. Inability to comply with protocol-specified hospitalization and restrictions
2. Richter's transformation
3. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other Infection (excluding Nail bed infection fungal) at study entry or any major Infection (as evaluated by the investigators) within 4 weeks prior to first study treatment Contacts and Locations
4. Suspected or Latent tuberculosis disease (confirmed by positive IFNγ release assay)
5. Positive test result for Chronic hepatitis B virus (HBV) Infection (defined as positive Hepatitis B surface antigen [HBsAg] serology).

   - Patients with occult or previous HBV Infection (defined as HBsAg negative and Hepatitis B core antibody [HBcAb] positive) may be included if HBV DNA is undetectable, provided they are willing to undergo HBV DNA testing monthly during study treatment (or on Day 1 of each cycle) and monthly for at least 12 months after the last cycle, and are willing to receive appropriate antiviral therapy.
6. Positive Hepatitis C virus (HCV) Antibody test

   - Patients with HCV Polymerase chain reaction are eligible only if the PCR (Antibody positive) is negative for HCV RNA.
7. Known HIV seropositive status

   - For patients with unknown HIV status, HIV testing will be performed at screening if required by local regulations.
8. Known or suspected chronic active Epstein-Barr Viral infection
9. Known or suspected history of Haemophagocytic lymphohistiocytosis (H LH)
10. Pregnancy or lactating, or planning to Pregnancy during treatment and for at least 3 months after the last dose of Gpt or within 2 months after the last dose of Glofitamab
11. A history of treatment-emergent Immunization related Immunization associated with prior Adverse event treatment agents as follows:

    * Grade 3 Adverse event, except for Grade 3 endocrinopathy managed with alternative therapy
    * Grade 1-2 Adverse event that did not return to baseline after Therapy cessation
12. Documented refractory to Obinutuzumab monotherapy
13. Active autoimmune disease requiring treatment requires investigator assessment of Immunization
14. Evidence of significant, uncontrolled concomitant disease that could affect adherence to the study protocol or interpretation of results, including Immunization, relevant Lung disorder history (Bronchospasm, Obstruction Pneumopathy), and known autoimmune Diabetes mellitus
15. History of severe Allergy or Allergic reaction to monoclonal antibody therapy (or recombinant antibody-associated fusion Protein)
16. History of confirmed progressive multifocal Leukoencephalopathy (PML)
17. Current or past history of CNS Lymphoma
18. Current or past history of CNS disease such as Stroke, Epilepsy, CNS Vasculitis, or neurodegenerative disease
19. Another invasive Neoplasm malignant within the last 2 years (except Basal cell carcinoma and Neoplasm with a low likelihood of recurrence)
20. Serious or extensive Angina unstable such as New York Heart disorder Association Class III or IV or objectively assessed Class C or D Cardiac disorder, Myocardial infarction within the last 6 months, unstable Arrhythmia, or Cardiovascular disorder
21. Administration of a live attenuated vaccine within 4 weeks prior to Gpt infusion, or anticipated need for a live attenuated vaccine during the study. ( Note: Flu vaccination should only be administered during the Flu season. Patients must not receive live attenuated Flu vaccine at any time during study treatment.)
22. Systemic Tumour necrosis agents (including but not limited to Cap Phosphorus amide, thiazolyl Purines, methotrexate, thalidomide, and anti Ammonia factor agents) within 2 weeks prior to Gpt infusions

    * Corticosteroid therapy with ≤ 25 mg/day prednisone or equivalent is allowed.
    * Inhaled and topical steroids are allowed.
23. History of illicit drugs or Alcohol abuse within 12 months prior to screening, as judged by the investigators.
24. Any other disease, metabolic dysfunction, Physical examination result, or clinical lab result reasonably suspecting a disease or condition that contraindicates the use of an investigational drug
25. Investigators should review the Vaccination status of potential study patients considered for this study and follow local disease control and prevention guidelines for vaccination of any other non-live vaccinated adults aiming to prevent infectious diseases prior to the study.
26. Any mental or Cognitive disorder that would limit the understanding, conduct, and compliance with the informed consent form;
27. Pregnancy or lactating females, or females or male partners planning to Pregnancy during the study;
28. Other situations that the investigators consider Discomfort to be eligible for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
complete response rate (CR) | up to the end of 12 cycles of treatment (each cycle is 28 days)
  To assess the complete response rate (CR) at the end of treatment with Glofitamab combination with chidamide.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to the end of 12 cycles of treatment (each cycle is 28 days)
  Objective Response Rate (ORR) is defined as the proportion of subjects who achieve CR or PR after treatment of Glofitamab combination with chidamide.
Duration of Response (DoR) | up to 2 years
  The length of time between the achievement of criteria for response to treatment (first documented complete or partial response) and the first documented relapse or progression.
Progression-free survival (PFS) | up to 2 years
  The time from the enrollment of a subject to the occurrence of (in any way) progression of disease or Death for any reason. patients with indeterminate recurrence or Death at the last follow-up, defined as the date of the last Investigation
OS | up to 2 years
  The time from subject enrollment to Death caused by any reason. for patients lost to follow-up, the time of the last follow-up; for patients still alive at the end of study, the date of the end of follow-up.

OTHER OUTCOMES:
To identify biomarkers | up to 2 years
  To identify biomarkers that may predict response to a combination regimen, biomarkers associated with progression to a more severe disease state, biomarkers that are sensitive to the development of Adverse event, biomarkers that provide evidence of the activity of the combination, or biomarkers that may enhance the understanding or understanding of the biology of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Insititute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No